CLINICAL TRIAL: NCT00378872
Title: Prospective Randomised Trial Comparing Intraoperative Topical Quixil and Intravenous Tranexamic Acid, in Reduction of Blood Loss Following Primary Hip & Knee Joint Replacement Surgery.
Brief Title: Tranexamic Acid vs. Quixil - Reducing Blood Loss in Joint Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Golden Jubilee National Hospital (Other Government)
Responsible Party: Mr Andrew Kinninmonth, Golden Jubilee National Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GJNH-06-01; Eudract number 2006-001299-19
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Hemorrhage; Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: IV Tranexamic acid 10mg/kg pt body weight
Drug: Quixil topical sealant

SUMMARY:
We will compare the effectiveness of Quixil and Tranexamic acid in reducing bleeding during hip and knee joint replacements.

DETAILED DESCRIPTION:
This is a prospective randomised controlled trial to compare the benefits of Quixil vs. Tranexamic acid in reducing blood loss.

Both medicines are used for the reduction of blood loss in major joint surgery; previous studies have shown each one to be effective and safe, but they have not been directly compared in this setting.

We will compare the blood loss in each of 3 groups: tranexamic acid used, Quixil used, and control group (neither drug used). Blood loss is to be calculated from height, body weight and difference between pre and post-operation haematocrit.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are to undergo elective hip or knee joint replacement
* Must be cemented arthroplasty
* Must be primary arthroplasty

Exclusion Criteria:

* Uncemented arthroplasty.
* Revision arthroplasty.
* Patients on anticoagulant (warfarin, low molecular weight heparin) or other medication known to affect clotting (except aspirin, which is to be given as part of standard DVT prophylaxis in all cases).
* Other drugs that may affect the activity of the drugs under investigation.
* Allergy to asprin (all patients to receive 150mg aspirin as standard DVT prophylaxis for 6 weeks).
* Patients with known coagulopathy (APTT or PT outside normal range pre-operatively).
* Previous reaction or ethical/religious objection to receiving blood products (Quixil contains a derivative of human blood).
* Pregnancy or breastfeeding.
* Patients who have a past medical history of thrombo-embolism at any time.
* Patients who need intravenous fluid administration for greater than 24 hours following operation.
* Patients who need allogenic blood transfusion within study period.
* Jehovah's Witnesses, or any other group of patients with ethical objections to receiving blood products.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Blood loss as calculated from change in haematocrit

CONTACTS AND LOCATIONS:
Overall Officials: Jamie S McConnell, MB BCh MRCS, Principal Investigator — Golden Jubilee National Hospital, NHS Scotland
Locations (1):
- Golden Jubilee National Hospital, Clydebank, Scotland, United Kingdom

REFERENCES:
- [Background] Benoni G, Fredin H. Fibrinolytic inhibition with tranexamic acid reduces blood loss and blood transfusion after knee arthroplasty: a prospective, randomised, double-blind study of 86 patients. J Bone Joint Surg Br. 1996 May;78(3):434-40. PMID 8636182
- [Background] Hiippala ST, Strid LJ, Wennerstrand MI, Arvela JV, Niemela HM, Mantyla SK, Kuisma RP, Ylinen JE. Tranexamic acid radically decreases blood loss and transfusions associated with total knee arthroplasty. Anesth Analg. 1997 Apr;84(4):839-44. doi: 10.1097/00000539-199704000-00026. PMID 9085968
- [Background] Ho KM, Ismail H. Use of intravenous tranexamic acid to reduce allogeneic blood transfusion in total hip and knee arthroplasty: a meta-analysis. Anaesth Intensive Care. 2003 Oct;31(5):529-37. doi: 10.1177/0310057X0303100507. PMID 14601276
- [Background] Husted H, Blond L, Sonne-Holm S, Holm G, Jacobsen TW, Gebuhr P. Tranexamic acid reduces blood loss and blood transfusions in primary total hip arthroplasty: a prospective randomized double-blind study in 40 patients. Acta Orthop Scand. 2003 Dec;74(6):665-9. doi: 10.1080/00016470310018171. PMID 14763696
- [Background] Levy O, Martinowitz U, Oran A, Tauber C, Horoszowski H. The use of fibrin tissue adhesive to reduce blood loss and the need for blood transfusion after total knee arthroplasty. A prospective, randomized, multicenter study. J Bone Joint Surg Am. 1999 Nov;81(11):1580-8. doi: 10.2106/00004623-199911000-00010. PMID 10565650
- [Background] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Background] Sehat KR, Evans RL, Newman JH. Hidden blood loss following hip and knee arthroplasty. Correct management of blood loss should take hidden loss into account. J Bone Joint Surg Br. 2004 May;86(4):561-5. PMID 15174554
- [Background] Wang GJ, Hungerford DS, Savory CG, Rosenberg AG, Mont MA, Burks SG, Mayers SL, Spotnitz WD. Use of fibrin sealant to reduce bloody drainage and hemoglobin loss after total knee arthroplasty: a brief note on a randomized prospective trial. J Bone Joint Surg Am. 2001 Oct;83(10):1503-5. doi: 10.2106/00004623-200110000-00007. PMID 11679600
- [Background] Zohar E, Fredman B, Ellis M, Luban I, Stern A, Jedeikin R. A comparative study of the postoperative allogeneic blood-sparing effect of tranexamic acid versus acute normovolemic hemodilution after total knee replacement. Anesth Analg. 1999 Dec;89(6):1382-7. doi: 10.1097/00000539-199912000-00010. PMID 10589612
- [Derived] McConnell JS, Shewale S, Munro NA, Shah K, Deakin AH, Kinninmonth AW. Reduction of blood loss in primary hip arthroplasty with tranexamic acid or fibrin spray. Acta Orthop. 2011 Dec;82(6):660-3. doi: 10.3109/17453674.2011.623568. Epub 2011 Oct 17. PMID 21999623
- [Derived] McConnell JS, Shewale S, Munro NA, Shah K, Deakin AH, Kinninmonth AW. Reducing blood loss in primary knee arthroplasty: a prospective randomised controlled trial of tranexamic acid and fibrin spray. Knee. 2012 Aug;19(4):295-8. doi: 10.1016/j.knee.2011.06.004. Epub 2011 Jul 5. PMID 21733697